CLINICAL TRIAL: NCT06663982
Title: Periosteal Inhibition Technique With Connective Tissue Graft and Leucocyte- Platelet Rich Fibrin in Alveolar Ridge Preservation: a Randomized Controlled Clinical Trial
Brief Title: Connective Tissue Graft and Leucocyte - Platelet Rich Fibrin in Alveolar Ridge Preservation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Michele Paolantonio, Full Professor, G. d'Annunzio University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27102024
Record Dates: First submitted 2024-10-27; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Alveolar Socket Preservation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CTG + L-PRF (Experimental)
  Interventions: Procedure: Connective tissue graft + L-PRF
- L-PRF (Active Comparator)
  Interventions: Procedure: L-PRF

INTERVENTIONS:
Procedure: Connective tissue graft + L-PRF — After administering local anesthesia, an atraumatic extraction will be conducted, preserving the buccal bone and carefully debriding the alveolar socket. Following papilla incisions, an intra-sulcular incision on the vestibular side of the extraction socket will be extended with a #15c scalpel, creating a socket to insert the connective tissue graft (CTG). The CTG will be harvested from the palatal area following a specific incision technique to obtain a graft around 1.5 mm thick, which will be fixed with a mattress suture.
  Then the socket will be filled with L-PRF plugs. A collagen sponge will cover the extraction socket and L-PRF, secured with a 4-0 cross suture. Sutures will be removed after 15 days.
  Arms: CTG + L-PRF
Procedure: L-PRF — After administering local anesthesia, an atraumatic extraction will be conducted, preserving the buccal bone and carefully debriding the alveolar socket.
  Then the socket will be filled with L-PRF plugs. A collagen sponge will cover the extraction socket and L-PRF, secured with a 4-0 cross suture. Sutures will be removed after 15 days.
  Arms: L-PRF

SUMMARY:
The purpose of our randomized controlled clinical trial is to evaluate radiographic bone dimensional changes and soft tissue healing and thickness after teeth extraction and the implementation of alveolar ridge preservation (RAP) procedures that will involve the application of L-PRF inside the socket in association with a connective tissue graft (CTG) used as a barrier with the periosteal inhibition technique (PI). The present experimental treatment (test group) will be compared with an active comparator (control group) which will involve the insertion of L-PRF alone inside the socket.

ELIGIBILITY:
* Age > 18 years old;
* General good health (ASA I-II);
* Adequate oral hygiene (Full Mouth Plaque Score ≤ 20%, Full Mouth Bleeding Score ≤ 20%);
* Presence of one or more hopeless teeth requiring extraction.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-12-09 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Horizontal Bone Crest | 4 months
  Horizontal width of the alveolar ridge

IPD SHARING:
Plan to Share IPD: Undecided